CLINICAL TRIAL: NCT06393738
Title: A Phase 1 First in Human Study of ARV-393 in Adult Participants With Advanced Non-Hodgkin's Lymphoma
Brief Title: A Study of ARV-393 in Relapsed/Refractory Non-Hodgkin Lymphoma.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Arvinas Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ARV-393-101; 2023-510136-36-00 (EU CTIS Number)
Record Dates: First submitted 2024-04-25; First posted 2024-05-01 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Relapsed/Refractory (R/R) Mature B Cell Non Hodgkin Lymphoma (NHL); Relapsed/Refractory (R/R) Angioimmunoblastic T-cell Lymphoma (AITL)
Keywords: Relapsed/Refractory B cell Non Hodgkin Lymphoma (NHL); Relapsed/Refractory Angioimmunoblastic T-cell lymphoma (AITL); Advanced non-Hodgkin Lymphoma; advanced NHL; relapsed non-Hodgkin Lymphoma; refractory non-Hodgkin Lymphoma; B Cell Advanced Non-Hodgkin Lymphoma
MeSH Terms: conditions — Recurrence; Immunoblastic Lymphadenopathy; Lymphoma, B-Cell; Lymphoma, Non-Hodgkin | interventions — glofitamab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A Monotherapy Dose escalation (Experimental): Participants with R/R NHL will receive ARV-393 dose escalation beginning at dose level 1
  Interventions: Drug: ARV-393
- Part B Monotherapy: Dose expansion/optimization (Experimental): Dose expansion and optimization of ARV-393 will be conducted in Part B to determine the recommended phase 2 dose (RP2D) for participants with R/R NHL
  Interventions: Drug: ARV-393
- Part C Combination therapy: Dose escalation (Experimental): Participants with R/R diffuse large B-cell lymphoma (DLBCL) will receive ARV-393 in combination with glofitamab, beginning at an ARV-393 dose informed by the Part A. Glofitamab will be given per labelled prescribing information. Part C will be conducted in non-USA centers.
  Interventions: Drug: ARV-393; Drug: Glofitamab
- Part D Combination therapy: Dose expansion/optimization (Experimental): Part D will be an optimization of ARV-393 in combination with glofitamab to determine a potential RP2D for ARV-393 in the combination regimen. Part D will be conducted in non-USA centers in participants with R/R DLBCL.
  Interventions: Drug: ARV-393; Drug: Glofitamab

INTERVENTIONS:
Drug: ARV-393 — Oral daily dose of ARV-393 at a specified dose level
Drug: Glofitamab — Glofitamab infusion per labelled prescribing information
  Arms: Part C Combination therapy: Dose escalation; Part D Combination therapy: Dose expansion/optimization

SUMMARY:
This clinical trial is studying the safety and potential anti-tumor activity of an investigational drug called ARV-393 in patients diagnosed with advanced Relapsed/Refractory non-Hodgkin's lymphoma (R/R NHL) to determine if ARV-393 may be a possible treatment option.

ARV-393 is thought to work by breaking down a protein present in many types of non-Hodgkins lymphomas, which may prevent, slow or stop tumor growth. This is the first time ARV-393 will be used by people. The investigational drug will be given as an oral tablet.

DETAILED DESCRIPTION:
This is an open-label, global, multi-center monotherapy and combination dose escalation and dose optimization study to evaluate safety, tolerability and preliminary efficacy of ARV-393. The study will evaluate the safety and tolerability in ascending doses of ARV-393 as monotherapy (A) and in combination with glofitamab (C), as well as determine the RP2D in the dose optimization parts (B for monotherapy) and in combination with glofitamab (D for combination therapy). The monotherapy portions of the study will include participants with R/R NHL. The combination therapy portions of the study with glofitamab will include participants with R/R DLBCL.

ELIGIBILITY:
Inclusion Criteria:

* For Part A and B: Have relapsed/refractory NHL and >=2 prior systemic therapies, (including rituximab), and be ineligible for known therapies with demonstrated clinical benefit per investigator assessment or, histologically confirmed AITL that has recurred or progressed following institutional standard of care therapy.
* For Part C and D: Have R/R DLBCL, not otherwise specified [NOS (DLBCL, NOS)] or large B-cell lymphoma (LBCL) arising from follicular lymphoma and have received two or more lines of systemic therapy.
* Have at least one bi dimensionally measurable lesion >1.5-centimeter (cm) in largest dimension for nodal or >1.0 cm for extranodal lesion.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1 (NOTE: For Part A only - ECOG PS of 2 is allowed for participants with secondary CNS lymphoma).
* Adequate bone marrow function
* Adequate kidney function
* Adequate Liver Function

Exclusion Criteria:

* Current or past history of peripheral eosinophilia, hypereosinophilic syndrome (HES), organ-specific eosinophilic disorder, or drug reaction with eosinophilia and systemic symptoms (DRESS).
* Prior allogeneic stem cell transplant (SCT) or solid organ transplantation.
* Any other active malignancy within 3 years prior to enrollment, except for adequately treated basal cell or squamous cell skin cancer, melanoma in situ or carcinoma in situ of the breast or cervix, and prostate cancer with active surveillance.
* Any of the following in the previous 6 months:

  * Myocardial infarction, long QT syndrome or family history of long QT syndrome, or Torsade de Pointes;
  * Clinically important atrial or ventricular arrhythmias;
  * Serious conduction system abnormalities, 3rd degree atrioventricular (AV block), unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure (CHF), New York Heart Association Class III or IV;
  * Cerebrovascular accident, transient ischemic attack, symptomatic pulmonary embolism, and/or other clinically significant episode of thromboembolic disease;
* Active inflammatory gastrointestinal (GI) disease, chronic diarrhea, previous gastric resection, or lap band surgery.
* Uncontrolled hypertension despite optimal medical treatment
* History of myocarditis.
* In ability to comply with listed prohibited treatments.
* Standard 12-lead electrocardiogram (ECG) that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results.
* Cardiac ejection fraction <45%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Estimated)
Dates: Start 2024-09-05 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities During First 28 Days | 28 days from first study dosing
  Percentage of participants in dose escalation arm at a given dose cohort with AEs meeting protocol defined dose limiting toxicities during cycle 1 (28 days)
Percentage of Participants With Adverse Events Characterized by Severity, Seriousness, and Relationship to Study Drug as a Measure of Safety and Tolerability | Parts A and B: From the study baseline to 30 days after last dose of ARV-393; Parts C and D: From the study baseline to 40 days after last dose of ARV-393
  Adverse events as characterized by type, frequency, severity, seriousness, and relationship to study drug
Number of Participants With Abnormal Vital Signs, Abnormal ECG Readings (QT Interval) and Abnormal Laboratory Parameters | Parts A and B: From the study baseline to 30 days after last dose of ARV-393; Parts C and D: From the study baseline to 40 days after last dose of ARV-393
  Shifts in vital signs, ECGs, and laboratory parameters from study baseline
Percentage of Participants With Grade 3 or Grade 4 Clinical Lab Abnormalities Using the Common Terminology Criteria for Adverse Events (CTCAE) With Scale From Grade 1 Grade 5. Higher Score Means Worse Outcome | Parts A and B: From the study baseline to 30 days after last dose of ARV-393; Parts C and D: From the study baseline to 40 days after last dose of ARV-393
  Incidence of Grade 3 and Grade 4 clinical laboratory abnormalities

SECONDARY OUTCOMES:
Area Under the Curve to the End of the Dosing Period (Auctau) for ARV-393 | 4 months from first drug dosing
  Assessment of pharmacokinetic parameter AUC
Area Under the Concentration Versus Time Curve, from 0 To Last Measurable Concentration (AUC0-Last) for ARV-393 | Time Frame: 4 months from first drug dosing
  Assessment of pharmacokinetic parameter AUC
Maximum Concentration (Cmax) for ARV-393 | 4 months from first drug dosing
  Cmax is an assessment of pharmacokinetic parameter
Minimum Concentration (Cmin) for ARV-393 | 4 months from first drug dosing
  Cmin is an assessment of pharmacokinetic parameter
Time to Maximum Concentration (Tmax) for ARV-393 | 4 months from first drug dosing
  Tmax is an assessment of pharmacokinetic parameter
Oral Clearance (CL/F) for ARV-393 | 4 months from first drug dosing
  CL/F is an assessment of pharmacokinetic parameter
Volume of Distribution (Vd/F) for ARV-393 | 4 months from first drug dosing
  Vd/F is a proportionality factor that relates the amount of drug in the body to the concentration of drug measured in a biological fluid.
Overall Response Rate (ORR) Based on Investigator Assessments of Response According to Lugano Response Criteria for NHL and International Primary Central Nervous System Lymphoma (PCNSL) Criteria for Central Nervous System (CNS Lymphoma), if Applicable | Approximately 2 years
  ORR is a parameter measuring the anti-tumor activity of the study intervention. It is the percentage of participants reaching a complete response or partial response to the study treatment.
Complete Response Rate (CRR) Based on Investigator Assessments of Response According to the Lugano Response Criteria for NHL and the International PCNSL Criteria for CNS Lymphoma, if Applicable | Approximately 2 years
  CRR is a parameter measuring the anti-tumor activity of the study intervention. CRR is percentage of participants with best of response reported as complete response.
Duration of Response (DOR) Based on Investigator Assessments of Response According to the Lugano Response Criteria for NHL and the International PCNSL Criteria for CNS Lymphoma, if Applicable | Approximately 2 years
  DOR is the time from the initial response (CR or PR) to the date of progression, or death, whichever occurs first. It is a parameter measuring the anti-tumor activity of the study intervention.

CONTACTS AND LOCATIONS:
Locations (16):
- United States (7):
  - Clinical Trial Site, New Haven, Connecticut
  - Clinical Trial Site, Detroit, Michigan
  - Clinical Trial Site, New Brunswick, New Jersey
  - Clinical Trial Site, New York, New York
  - Clinical Trial Site, Cleveland, Ohio
  - Clinical Trial Site, Nashville, Tennessee
  - Clinical Trial Site, Houston, Texas
- Canada (2):
  - Clinical Trial Site, Toronto, Ontario
  - Clinical Trial Site, Montreal, Quebec
- Denmark (2):
  - Clinical Trial Site, Copenhagen
  - Clinical Trial Site, Odense C
- Spain (5):
  - Clinical Trial Site, El Palmar, Murcia
  - Clinical Trial Site, Pamplona, Navarre
  - Clinical Trial Site, Barcelona
  - Clinical Trial Site, Madrid
  - Clinical Trial Site, Salamanca

IPD SHARING:
Plan to Share IPD: No